CLINICAL TRIAL: NCT06911944
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 4 Dose-Escalation Study Evaluating the Safety, Tolerability, and Efficacy of Donanemab in Adults With Down Syndrome
Brief Title: Amyloid Lowering for Alzheimer's in Down's With Donanemab Investigation
Acronym: ALADDIN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Rafii, MD, PhD (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Eli Lilly and Company (Industry); Alzheimer's Clinical Trials Consortium (Other); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Sponsor-Investigator, Michael Rafii, MD, PhD, Medical Director of the Alzheimer's Therapeutic Research Institute (ATRI) and Professor of Clinical Neurology at the Keck School of Medicine, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATRI-016; 5R33AG066543 (NIH)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Down Syndrome (DS); Down Syndrome (Trisomy 21); Alzheimer Disease; Amyloid Beta Protein
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease; Plaque, Amyloid | interventions — donanemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- donanemab (Experimental): Donanemab will be administered per label instructions and the pharmacy manual as an IV infusion every 4 weeks using an up-titration regimen that will allow participants to reach a target dose of 1400 mg within 12 weeks
  Interventions: Drug: Donanemab
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donanemab — Donanemab will be administered as an IV infusion every 4 weeks using an up-titration regimen that will allow participants to reach a target dose of 1400 mg within 24 weeks.
  Other Names: Kisunla
  Arms: donanemab
Drug: Placebo — The control product (placebo) will be supplied in vials containing 350 mg/20 mL of donanemab Placebo for donanemab is supplied to the clinical site to match the active study intervention and contains only inactive ingredients. Normal sterile saline solution (0.9% sodium chloride) will be used for dilution.
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn if donanemab can reduce levels of amyloid in the brain, and if donanemab is safe and well-tolerated in participants with Down syndrome.

The main questions it aims to answer are: Does donanemab reduce amyloid in the brain? Is donanemab safe and well-tolerated in people with Down syndrome? Researchers will compare donanemab to a placebo (a look-alike substance that contains no drug) to see if donanemab works to reduce levels of amyloid in the brain.

Participants in the study will be 35-50 years old and will be in the study for 12 months. Participants will then stay in the study for an additional 12 months in an long-term extension where all participants will receive donanemab. Participants who had a reduction in amyloid (measured by amyloid brain scan) by the end of the first 12 months will receive placebo for the long-term extension, while participants who did not have an amyloid reduction will receive study donanemab for the long-term extension. Everyone (participants and study staff) will remain blinded to treatment for the duration of the study.

Participants will:

* Have intravenous (IV) infusions of donanemab (or placebo) every 4 weeks
* Visit the clinic once every other month for checkups and tests. These tests will include brain scans (magnetic resonance imaging [MRI] and positron emission tomography [PET] ), blood draws and memory tests.
* Have a study partner who who can provide information about the participant and can join participant for some of the study visits.

DETAILED DESCRIPTION:
The conduct of this Phase 4 clinical study is intended to evaluate the effect of donanemab, a humanized monoclonal antibody, on brain amyloid (centiloids), in the non-demented DS population, with the primary objective of reducing amyloid accumulation. Concurrently, the study aims to investigate the safety and tolerability, and therapeutic potential of donanemab while maintaining the safety and tolerability observed in clinical studies in early AD populations up to the dose of 1400mg.

Safety, tolerability, and efficacy of donanemab will be assessed in a non-demented DS population in the range of 35-50 years of age who are cognitively stable or have Mild Cognitive Impairment (MCI), which could indicate preclinical and prodromal AD, in a genetic population with ≥18 centiloids on amyloid-PET.

The study will have a duration of approximately 12 months (52 weeks). A long-term extension (LTE) will also be included, lasting an additional 12 months (52 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of the participant's informed consent to study procedures
2. Ages 35-50 years (inclusive).
3. Plasma Phosphorylated tau (pTau) 217 levels at screening consistent with amyloid PET eligibility.
4. Diagnosis of Down syndrome (including trisomy 21, mosaic trisomy 21, Robertsonian translocation trisomy 21, or partial trisomy 21) as confirmed by medical record review or Karyotype genetic testing.
5. Intelligence quotient (IQ) equal to or greater than 40 based on Kaufman Brief Intelligence Test, Second Edition.
6. Participants must be in good general health as evidenced by medical history with no diagnosis of dementia.
7. Elevated brain amyloid (>18 centiloids) at screening.
8. Stable dose of permitted medications as described protocol for 4 weeks prior to screening.
9. In the opinion of the site PI, has a study partner able and willing to provide accurate information (including clinical symptoms and medical history) about the participant and participate in study visits and informant-based assessments (usually requires at least 5 hours of contact per week) for the duration of the study.
10. As assessed by the site PI, participant is likely to be able to comply with the protocol for the duration of the study, and has adequate vision, hearing (hearing aid permitted), and literacy sufficient for compliance with required testing procedures.
11. Must complete all screening evaluations as outlined in protocol

Exclusion Criteria:

1. Females who are lactating or pregnant (as confirmed by a urine pregnancy test) during screening, or plan to become pregnant during the study.
2. Females of childbearing potential or males with a female partner of childbearing potential who did not use a highly effective method of contraception within 28 days of screening alongside with a suitable barrier method (e.g., male condom) and/or are not willing to use both methods for the duration of their participation in the study and for 3 months after the last dose of study drug.
3. Weight less than 40kg at screening.
4. Lack of good venous access such that intravenous (IV) drug delivery or multiple blood draws would be precluded.
5. Suspected or known allergic reactions, adverse reactions, or hypersensitivity to humanized monoclonal antibodies or any components of the study treatments (donanemab or placebo).
6. Previous treatment with donanemab unless there is firm evidence that the participant received placebo only.
7. Prior or current treatment with a prohibited medication as described in protocol.
8. Enrollment in another investigational study, or intake of investigational drug, within 30 days prior to screening or five half-lives of the investigational drug, whichever is longer.
9. MRI scan at screening showing a single area of cerebral vasogenic edema, superficial siderosis, or evidence of a prior macro-hemorrhage, or showing more than one (1) cerebral microhemorrhage (regardless of their anatomical location with a diagnostic characterization as "definite"), evidence of space occupying lesions, more than two (2) lacunar infarcts, or one (1) infarct larger than 1cm in diameter, severe white matter disease, and structural evidence of alternative pathology not consistent with AD and considered to be at the origin of participant's symptoms.

   NOTE: Small incidental meningiomas and arachnoid cysts (<1cm in diameter) may be permitted with Medical Monitor review and approval.
10. Contraindication(s) to MRI studies, including metal (ferromagnetic) implants, a cardiac pacemaker or other devices that are not compatible with MRI, and/or severe claustrophobia.
11. Contraindications to amyloid positron emission tomography (PET) imaging and/or use of florbetapir.
12. Any unstable and/or clinically significant medical condition likely to hamper the evaluation of safety and/or efficacy of study drug (e.g., moderate and/or severe untreated obstructive sleep apnea, clinically significant reduction in serum B12 or folate levels, clinically significant abnormalities of thyroid function, stroke, or other cerebrovascular conditions), as per the site PI's judgement.
13. History of severe allergic reaction (e.g., anaphylaxis) including, but not limited to: severe allergic reaction to previous vaccines, foods, and/or medications.
14. Hospitalization within 30 days prior to screening or baseline.
15. Clinically significant infections or major surgical operation within 3 months prior to screening.
16. History of chronic or recurrent infections judged to be clinically significant by the site PI and which would potentially hamper the evaluation of efficacy and safety assessments.
17. Myocardial infarction within one (1) year prior to baseline, unstable angina pectoris, or significant coronary artery disease.
18. History of cancer within the past five (5) years other than treated squamous cell carcinoma, basal cell carcinoma and melanoma in-situ, in-situ prostate cancer, or in-situ breast cancer, which have been fully removed and are considered cured.
19. History or presence of immunological or inflammatory conditions, including neurological disorders, judged to be clinically significant by the site PI.
20. History of meningitis or meningoencephalitis.
21. History of moderate or severe traumatic brain injury.
22. History or presence of uncontrolled seizures. If history of seizures, they must be well controlled with no occurrence of seizures in the 2 years prior to study screening. The use of antiepileptic medications is permitted.
23. Concomitant or past history of psychiatric or neurologic disorder (e.g., head injury with loss of consciousness, symptomatic stroke, Parkinson's disease, severe carotid occlusive disease, transient ischemic attacks, hemorrhagic and/or non-hemorrhagic stroke) other than those considered to be related to AD.
24. Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for drug or alcohol abuse or dependence currently met within the past 5 years.
25. Significant risk of suicide defined, using the Columbia-Suicide Severity Rating Scale (C-SSRS) (Child Version), as the participant answering "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behavior within the past 12 months.
26. Clinically significant abnormal vital signs including sustained sitting blood pressure >160/90 millimeters of mercury (mmHg).
27. Participants with diabetes mellitus with hemoglobin A1c (HbA1c) levels of ≥8.0%.
28. In the opinion of the site PI, clinically significant deviations from normal values for hematologic parameters, liver function tests, and other biochemical measures.
29. Participants with a known history of human immunodeficiency virus (HIV-1 and 2).
30. Participants with known history of acute/chronic hepatitis B or C.
31. Clinically significant arrhythmias or other clinically significant abnormalities on electrocardiogram (ECG) at screening (minor abnormalities documented as clinically insignificant by the site PI are allowed).
32. Residing in a continuous care nursing facility.
33. For participants undergoing Lumbar Puncture (LP) as part of the optional longitudinal cerebrospinal fluid (CSF) biomarker sub-study, any contraindication to LP including, but not limited to: inability to tolerate an appropriately flexed position for the time necessary to perform an LP; international normalized ratio (INR) >1.4 or other metrics indicating coagulopathy; platelet count of <120,000/microliter(μL); infection at the desired lumbar puncture site; taking anti-coagulant medication within 90 days of LP (Note: low dose (up to 81 milligram (mg)) aspirin is permitted); degenerative arthritis of the lumbar spine; suspected or known non-communicating hydrocephalus or intracranial mass, or elevated intracranial pressure from any cause; prior history of spinal mass or trauma.
34. Participants unwilling to learn their APOE genotype and/or amyloid PET scan results
35. Participants who are apolipoprotein E ε4 (APOE ε4) homozygotes.
36. Participants who receive anti-coagulants or thrombolytics within 30 days prior to baseline. Any use of anticoagulants or thrombolytics during the study will lead to discontinuation of the study drug.
37. Participants with clotting disorders.
38. Any condition, which in the opinion of the site PI, Coordinating Center, regulatory sponsor, or Project Lead/Protocol PI, makes the participant unsuitable for inclusion.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on brain amyloid levels | 12 months
  Change in brain amyloid measured by amyloid PET imaging (amyloid centiloid levels) from baseline to 12 months. An increase indicates a worsening.

SECONDARY OUTCOMES:
Change from baseline to 12 months in the Modified Cued Recall Test (mCRT) | From baseline to 12 months
  The Modified Cued Recall Test (mCRT) is a cognitive assessment tool designed to evaluate memory and has been modified from a version developed for adults from the typical population. 12 items are presented for learning, 4 at a time, with each item accompanied by a unique category cue. The testing phase consists of 3 trials. Each trial begins with free recall of the test items; following free recall, a category cue is provided for those items not spontaneously recalled. Two scores are generated from the test, a Free Recall Score and a Total Score. A higher score indicates a better outcome.
Change from baseline in whole brain volume | From baseline to 12 months
  Change in whole brain volume as measured by MRI. A decrease indicates a worsening.
Change from baseline in brain hippocampal volume | From baseline to 12 months
  Change in brain hippocampal volume as measured by MRI. A decrease indicates a worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rafii, MD, PhD, Principal Investigator — University of Southern California (USC) Keck School of Medicine, Alzheimer's Therapeutic Research Institute (ATRI)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- See also: Alzheimer's Clinical Trials Consortium - Down Syndrome — https://www.actc-ds.org/